CLINICAL TRIAL: NCT02914730
Title: Insulin Dosing Practices in Persons With Diabetes on Multiple Daily Injections
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Medha Munshi, Director of Joslin Geriatric Diabetes Programs Beth Israel Deaconess Medical Center Associate Professor of Medicine, Harvard Medical School, Joslin Diabetes Center
Other Study IDs: CHS #2015-47
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Diabetes; Medication Adherence; Technology; Insulin
Keywords: diabetes; insulin; medication adherence
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
In this cross-sectional study the investigators will examine two populations: young adults with (ages 18-35) and older adults (ages 65 and over) with diabetes who are on > 2 insulin injections per day. The sample size for this observational study will be up to 125 patients. The investigators will issue a Common Sensing GoCap bluetooth-enabled pen cap that fits on the end of Solostar Lantus and Apidra insulin pens; this pen cap registers the position of the insulin pen plunger and automatically sends confirmation of dose delivery to a smartphone app.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes or insulin-requiring Type 2 diabetes
* > 2 insulin injections
* Age 18-35 or older than 65 years
* Use of glargine insulin as basal insulin
* Stable insulin doses for past 3 months

Exclusion Criteria:

* Previous tape/adhesive allergies with CGM sensors
* Visual or cognitive impairment with inability to self-administer insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this cross-sectional study the investigators will examine two populations: young adults with (ages 18-35) and older adults (ages 65 and over) with diabetes who are on > 2 insulin injections per day. The sample size for this observational study will be up to 125 patients.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Number of Missed Insulin Doses | 4 week use of blue tooth pen cap

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin DIabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Munshi MN, Slyne C, Greenberg JM, Greaves T, Lee A, Carl S, Atakov-Castillo A, Toschi E. Nonadherence to Insulin Therapy Detected by Bluetooth-Enabled Pen Cap Is Associated With Poor Glycemic Control. Diabetes Care. 2019 Jun;42(6):1129-1131. doi: 10.2337/dc18-1631. Epub 2019 Mar 12. PMID 30862650